CLINICAL TRIAL: NCT04528849
Title: Comparison of Ovulation Induction Cycle Outcomes Between Early and Late Dose Increments for Low Dose Gonadotropin Step-up Protocol Among Infertile Women Diagnosed With Polycystic Ovary Syndrome: Prospective Randomised Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Serkan Kahyaoglu, Associate Professor, M.D, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E1-20-377
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Polycystic Ovary Syndrome; Infertility, Female
Keywords: Polycystic ovary syndrome; Infertility; Low dose step-up; Gonadotropin; Ovulation induction
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility, Female; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early dose increment (Active Comparator): Patients who have received 25 IU gonadotropin dose increment on 7th day of ovulation induction
  Interventions: Drug: Gonadotropin dose increment timing
- Late dose increment (Active Comparator): Patients who have received 25 IU gonadotropin dose increment on 14th day of ovulation induction
  Interventions: Drug: Gonadotropin dose increment timing

INTERVENTIONS:
Drug: Gonadotropin dose increment timing — Gonadotropin dose increments of 25 IU will be utilized on 7th and 14th day of ovulation induction for each study group.

SUMMARY:
Low dose gonadotropin step-up ovulation induction treatment is the universally accepted and utilized teratment protocol for infertile women diagnosed with polycystic ovary syndrome (PCOS). First dose increment is advised on 14th day of ovarian stimulation with gonadotropins to decrease multiple follicle generation and cycle cancellation rates. However, clinicians impatiently increase gonadotropin dose on 7th day of stimulation without strong scientific evidence. This randomised controlled study will be the first study which will compare safety and ovulation induction cyle outcomes of early and late dose increments among infertile women diagnosed with PCOS.

DETAILED DESCRIPTION:
Low dose gonadotropin step-up ovulation induction treatment is the universally accepted and utilized teratment protocol for infertile women diagnosed with polycystic ovary syndrome. First dose increment is advised on 14th day of ovarian stimulation with gonadotropins to decrease multiple follicle generation and cycle cancellation rates. However, clinicians impatiently increase gonadotropin dose on 7th day of stimulation without strong scientific evidence. This randomised controlled study will be the first study which will compare safety and ovulation induction cyle outcomes of early and late dose increments among infertile women diagnosed with polycystic ovary syndrome.

We will start low dose step-up ovulation induction treatment by using 50 IU recombinant FSH for 21-39 years old non- obese patients (BMI <30 kg/m2) diagnosed with PCOS and . We will perform folliculometry on 7th day of ovulation induction. In case of absence for at least one >10 mm dominant follicle, we will randomise these women by using blind envelope selection method for assignment of early or late dose incerement groups. Half of the patients will receive 25 IU dose increment on 7th day of ovulation induction, remaining half will receive dose increment on 14th day of ovulation induction. We will continue ovarian stimulation without any other dose increment until 35th day of stimulation as deadline time restriction. We will perform folliculometry and serum estradiol measurement intermittently during ovulation induction. We will record ovulation induction cycle outcomes and clinical pregnancy results of the study group following finalization for treatment cyle of each patient. We will compare ovulation induction cycle outcomes of these two dose increment groups.

ELIGIBILITY:
Inclusion Criteria:Infertile women who have been diagnosed with PCOS based on Rotterdam criteriae and who have not succeeded to get pregnant by using oral ovulation induction agents and whose BMI levels are <30 kg/m2 will be included to the study.

Exclusion Criteria:Infertile women with tubal diseases, male factor infertility, endometriosis, previous pelvic surgery history, chronic systemic disease, BMI levels>30 kg/m2 and who are not voluntary to attend to the study will be excluded from the study.

Ages: 21 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-08-20 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2022-08-20 (Estimated)

PRIMARY OUTCOMES:
Number of preovulatory follicles | 35 days
  Number of >14 mm sized follicles at the end of the ovulation induction treatment

SECONDARY OUTCOMES:
Biochemical pregnancy rate | 2 weeks after ovulation triggering
  Serum pregnancy test will be performed 2 weeks after ovulation triggering
Clinical pregnancy rate | 3 weeks after ovulation triggering
  Clinical pregnancy rate which will be evaluated 3 weeks after ovulation triggering
Cycle length in days | 7-35 days
  Total number of ovulation induction days until ovulation triggering
Cycle cancellation | 35 days
  Cycle cancellation due to >=3 preovulatory follicles (>14 mm in size) at the end of the ovulation induction treatment
Multiple pregnancy rate | 3 weeks after ovulation triggering
  Multiple pregnancy rate which will be evaluated 3 weeks after ovulation triggering

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Kahyaoglu, M.D, Principal Investigator — Ankara City Hospital, Department of Reproductive Endocrinology
Locations (1):
- University of Health Sciences, Ankara City Hospital, Department of Reproductive Endocrinology, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Improved monofollicular ovulation in anovulatory or oligo-ovulatory women after a low-dose step-up protocol with weekly increments of 25 international units of follicle-stimulating hormone — https://pubmed.ncbi.nlm.nih.gov/16759926/
- See also: Pilot study of the optimal protocol of low dose step-up follicle stimulating hormone therapy for infertile women — https://pubmed.ncbi.nlm.nih.gov/30013434/
- See also: Ovulation induction with a starting dose of 50 IU of recombinant follicle stimulating hormone in WHO group II anovulatory women: the IO-50 study, a prospective, observational, multicentre, open trial — https://pubmed.ncbi.nlm.nih.gov/14664878/